CLINICAL TRIAL: NCT05172609
Title: An Exposure-Based Implementation Strategy to Decrease Clinician Anxiety About Delivering Suicide Prevention Evidence-Based Practices
Brief Title: An Exposure-Based Implementation Strategy to Decrease Clinician Anxiety Around Suicide Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 356336
Record Dates: First submitted 2021-08-25; First posted 2021-12-29 (Actual); Results first posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-07

CONDITIONS: Implementation Science

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure Based Implementation Strategy (EBIS) (Experimental): EBIS is informed by the latest science in exposure theory, borrowing heavily from brief exposure-based treatments that can be delivered in a single session. We anticipate that EBIS will occur in four phases that map on to standard exposure therapy practice for patients with anxiety disorders: psychoeducation, assessment, practice, and relapse prevention; however, the final version will depend on the outcomes of the preparatory phases of this study. Clinicians assigned to the EBIS arm will also receive all elements of IAU.
  Interventions: Behavioral: Exposure Based Implementation Strategy (EBIS)
- Implementation as Usual (IAU) (Active Comparator): Gold-standard IAU for SSAIs typically comprises pre-implementation preparation, didactic training, knowledge tests, experiential role plays, ongoing expert consultation, and providing certification status to clinicians who attain established benchmarks. Pre-implementation preparation will include provision of materials. Didactic training will occur in two parts: (1) suicide screening and assessment, and (2) Safety Planning Intervention (SPI) use. Part one will consist of materials we previously developed based on community clinician feedback. Part two will follow established SPI guidelines, including didactic training about SPI rationale and evidence base and experiential practice. IAU also will include supports for electronic health record integration (e.g., previously developed templates). After training, clinicians will receive 8 weeks of expert consultation to discuss implementation barriers and receive more role play practice.
  Interventions: Behavioral: Implementation as Usual (IAU)

INTERVENTIONS:
Behavioral: Exposure Based Implementation Strategy (EBIS) — EBIS will include psychoeducation, assessment/hierarchy building. guided practice, and guidance for application to clinical practice.
  Arms: Exposure Based Implementation Strategy (EBIS)
Behavioral: Implementation as Usual (IAU) — IAU will consist of standard didactic training and ongoing consultation activities for enrolled clinicians
  Arms: Implementation as Usual (IAU)

SUMMARY:
Study objectives are to design and pilot test a novel, exposure-based implementation strategy (EBIS) directly targeting clinician anxiety and low self-efficacy for use of evidence-based suicide screening, assessment, and intervention (SSAI) strategies with patients at risk for suicide in community settings. Early phases of this study will develop the EBIS in partnership with community clinicians (n = 15). The last phase of this study is a pilot clinical trial in which 40 community mental health clinicians will be randomized to receive either implementation as usual (IAU) or IAU+EBIS.

DETAILED DESCRIPTION:
This exploratory project brings together an interdisciplinary team to design and pilot-test an exposure-based implementation strategy (EBIS) to target clinician-level anxiety about suicide screening, assessment, and intervention (SSAI) use. We will test the effect of EBIS as an implementation strategy to augment Implementation as Usual (IAU) to enhance SSAI implementation in community mental health settings. Specifically, this study first will use participatory design methods to develop and refine EBIS in collaboration with a stakeholder advisory board of clinicians, administrators, and content experts. This study then will further iteratively refine EBIS with up to 15 clinicians in a pilot field test, using rapid cycle prototyping, in collaboration with the INSPIRE Methods Core. Clinicians in Aim 2 will also provide qualitative feedback on EBIS' ability to mitigate anxiety and increase self-efficacy to deliver SSAIs to optimize our ability to engage target mechanisms of clinician anxiety. In the final phase, this study will test the refined EBIS in a pilot implementation trial in which 40 community mental health clinicians will be randomized to receive either IAU or EBIS+IAU. Primary clinical trial dependent variables are EBIS acceptability and feasibility, measured through questionnaires, interviews, and recruitment and retention statistics; this pilot trial is not intended to be powered to detect effects. Secondary outcomes are preliminary effectiveness of EBIS on clinician-level implementation outcomes (SSAI adoption), and engagement of target implementation mechanisms (clinician anxiety and self-efficacy related to SSAI use), assessed via mixed methods.

Aim 1 did not include data collection from study participants. Activities in this aim only included refinement with the advisory board members who were not considered study participants.

Data collected in Aim 2 was largely descriptive and qualitative to inform EBIS development and refinement activities.

We are reporting Aim 3 data which included pilot randomization with clinicians. Data was collected at the following timepoints: Time 1: baseline measures completed before the training; Time 2: immediately after completing the training; Time 3: two weeks after completing the training; Time 4: 12 weeks after completing the training.

ELIGIBILITY:
Inclusion Criteria:

* Practicing mental health clinicians who provide direct mental health services to a treatment-seeking population
* Proficient in the English language
* Have access to a computer with internet connectivity

Exclusion Criteria:

* Participants will be excluded if they do not see any mental health patients that are at risk for suicide (e.g., they screen out high-risk patients for their individual practice).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania Department of Psychiatry, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Becker-Haimes EM, Brady M, Jamison J, Jager-Hyman S, Reilly ME, Patel E, Brown GK, Mandell DS, Oquendo MA. An exposure-based implementation strategy to decrease clinician anxiety about implementing suicide prevention evidence-based practices: protocol for development and pilot testing (Project CALMER). Implement Sci Commun. 2023 Nov 24;4(1):148. doi: 10.1186/s43058-023-00530-3. PMID 38001478

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We are reporting Aim 3 data which included pilot randomization with clinicians. Data from Aims 1 and 2 are not included as these aims were largely preparatory. Aim 3 data was collected at baseline before the training (Time 1), after the training (Time 2), two weeks after the training (Time 3), and 12 weeks after the training (Time 4). These clinician participants were recruited from 5 agencies between July to August 2023.
Pre-assignment Details: 42 participants were consented into the study. 3 dropped out before completing any study activities due to time constraints or a change in eligibility status. 39 completed baseline measures before randomization (time 1). Of the 39, 3 dropped out due to timing constraints or change in eligibility status. 36 were randomized to condition by training type.
Groups:
- Exposure Based Implementation Strategy (EBIS): EBIS is informed by the latest science in exposure theory, borrowing heavily from brief exposure-based treatments that can be delivered in a single session. EBIS occurred in four phases that map on to standard exposure therapy practice for patients with anxiety disorders: psychoeducation, assessment, practice, and relapse prevention. Clinicians assigned to the EBIS arm received all elements of the EBIS plus all elements of IAU.
  Exposure Based Implementation Strategy (EBIS): EBIS included psychoeducation, assessment/hierarchy building. guided practice, and guidance for application to clinical practice.
- Implementation as Usual (IAU): Gold-standard IAU for suicide screening, assessing, and intervening (SSAIs) typically comprises pre-implementation preparation, didactic training, knowledge tests, experiential role plays, ongoing expert consultation, and providing certification status to clinicians who attain established benchmarks. Pre-implementation preparation included provision of materials. Didactic training occurred in two parts: (1) suicide screening and assessment, and (2) Safety Planning Intervention (SPI) use. Part one consisted of materials we previously developed based on community clinician feedback. Part two followed established SPI guidelines, including didactic training about SPI rationale and evidence base and experiential practice. IAU also included supports for electronic health record integration (e.g., previously developed templates). After training, clinicians received 6 hours of expert consultation in small groups over 12 weeks to discuss implementation barriers and receive more role play practice.
  Implementation as Usual (IAU): IAU consisted of standard didactic training and ongoing consultation activities for enrolled clinicians
Period: Time 2
Arm/Group | Exposure Based Implementation Strategy (EBIS) | Implementation as Usual (IAU)
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Time 3
Arm/Group | Exposure Based Implementation Strategy (EBIS) | Implementation as Usual (IAU)
Started | 18 | 18
Completed | 17 | 17
Not Completed | 1 | 1
Not completed — Elected not to continue with study due to time constraints | 1 | 1
Period: Time 4
Arm/Group | Exposure Based Implementation Strategy (EBIS) | Implementation as Usual (IAU)
Started | 17 | 17
Completed | 16 | 16
Not Completed | 1 | 1
Not completed — Elected not to continue with study due to personal reasons unrelated to the study | 1 | 0
Not completed — Elected not to continue with study due to time constraints | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were captured from participants before randomization
Groups:
- Enrolled, Not Yet Randomized: Participant information reported below include Aim 3 data captured before participants were randomized into EBIS or IAU conditions. After participants consented to study participation, they completed baseline measures. Participants were randomized after all participants were consented 1:1 by training date (EBIS or IAU).
Arm/Group | Enrolled, Not Yet Randomized
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.0 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 23
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 42

OUTCOME MEASURES:

1. Primary Outcome: Clinician Perception of EBIS Acceptability for Clinical Practice at Time 4, 12 Weeks After Completing Training
Description: Acceptability of EBIS was measured with the Acceptability of Intervention Measure (AIM), a 4-item, psychometrically-validated measure that indexes the extent to which stakeholders believe an implementation strategy is acceptable. Items on the AIM are rated on a 5-point Likert scale (Range = 4-20) and higher scores indicate greater acceptability.
Time Frame: Time 4: 12 weeks after completing training
Population: After completing baseline measures, participants were randomized to training condition. By the end of the 12 week trial, 2 participants had dropped out of each study condition (n = 4).
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Implementation as Usual (IAU): Gold-standard IAU for SSAIs typically comprises pre-implementation preparation, didactic training, knowledge tests, experiential role plays, ongoing expert consultation, and providing certification status to clinicians who attain established benchmarks. Pre-implementation preparation included provision of materials. Didactic training occurred in two parts: (1) suicide screening and assessment, and (2) Safety Planning Intervention (SPI) use. Part one consisted of materials we previously developed based on community clinician feedback. Part two followed established SPI guidelines, including didactic training about SPI rationale and evidence base and experiential practice. IAU also included supports for electronic health record integration (e.g., previously developed templates). After training, clinicians received 6 hours of expert consultation in small groups over 12 weeks to discuss implementation barriers and receive more role play practice.
  Implementation as Usual (IAU): IAU consisted of standard didactic training and ongoing consultation activities for enrolled clinicians
Arm/Group | Exposure Based Implementation Strategy (EBIS) | Implementation as Usual (IAU)
Number analyzed (Participants) | 16 | 16
units on a scale | 4.55 (.53) | 4.56 (.46)
Statistical Analysis 1: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); T-tests between EBIS and IAU conditions at 12-week follow up for AIM; Test type: Equivalence — Margin difference of 1 standard deviation (SD) or higher was considered evidence of non-equivalence comparison; p = .47, t-test, 2 sided

2. Primary Outcome: Clinician Perception of EBIS Feasibility and Utility for Clinical Practice at Time 4, 12 Weeks After Completing Training
Description: Feasibility of EBIS was measured with the Feasibility of Intervention Measure (FIM), a 4-item measure that indexes the extent to which an implementation strategy is perceived as feasible. Items on the FIM are rated on a 5-point Likert scale (Range = 4-20) and higher scores indicate greater acceptability.
Time Frame: Time 4: 12 weeks after completing training
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure Based Implementation Strategy (EBIS) | Implementation as Usual (IAU)
Number analyzed (Participants) | 16 | 16
units on a scale | 4.59 (.48) | 4.63 (.47)
Statistical Analysis 1: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); T-tests between EBIS and IAU conditions at 12-week follow up for FIM; Test type: Equivalence — Margin difference of 1 SD or higher was considered evidence of non-equivalence comparison; p = .88, t-test, 2 sided

3. Secondary Outcome: Clinician Anxiety at 4 Timepoints Across 12 Weeks
Description: Clinician anxiety was assessed via 10-point Subjective Units of Distress (SUDS), a 10-point Likert rating of subjective distress where 1 = Not at all Distressed and 10 = Very Distressed. Clinicians rated their anxiety on screening and safety planning separately.
Time Frame: Time 1: baseline measures completed before the training; Time 2: immediately after completing the training; Time 3: two weeks after completing the training; Time 4: 12 weeks after completing the training.
Population: This measure was completed across four timepoints. 2 participants dropped out of the study after post-intervention measures. 2 additional participants dropped out after two week follow up measures
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure Based Implementation Strategy (EBIS) | Implementation as Usual (IAU)
Number analyzed (Participants) | 18 | 18
units on a scale
  Time 1: SUDS, screening | 4.28 (1.78) | 3.94 (2.36)
  Time 1: SUDS, planning | 4.67 (2.30) | 4.28 (2.11)
  Time 2: SUDS, screening | 5.06 (2.01) | 3.94 (2.29)
  Time 2: SUDS, planning | 5.50 (2.38) | 4.33 (2.97)
  Time 3: SUDS, screening: number analyzed (Participants) | 17 | 17
  Time 3: SUDS, screening | 4.59 (2.00) | 4.06 (2.14)
  Time 3: SUDS, planning: number analyzed (Participants) | 17 | 17
  Time 3: SUDS, planning | 4.76 (2.11) | 4.29 (2.57)
  Time 4: SUDS, screening: number analyzed (Participants) | 16 | 16
  Time 4: SUDS, screening | 3.75 (1.53) | 3.25 (1.77)
  Time 4: SUDS, planning: number analyzed (Participants) | 16 | 16
  Time 4: SUDS, planning | 3.50 (1.79) | 3.81 (2.43)
Statistical Analysis 1: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing SUDS screening rating at Time 3: two weeks after completing the training; Test type: Superiority; p = .46, t-test, 2 sided
Statistical Analysis 2: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing SUDS screening rating at Time 4: 12 weeks after completing the training; Test type: Superiority; p = .40, t-test, 2 sided
Statistical Analysis 3: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing SUDS planning rating at Time 3: two weeks after completing the training; Test type: Superiority; p = .56, t-test, 2 sided
Statistical Analysis 4: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing SUDS planning rating at Time 4: 12 weeks after completing the training; Test type: Superiority; p = .68, t-test, 2 sided
Statistical Analysis 5: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Repeated measures analysis of covariance (ANCOVA), controlling for organization: SUDS screening at timepoints 1, 3, and 4; Test type: Superiority; p = .87, ANCOVA
Statistical Analysis 6: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); repeated measures analysis of covariance (ANCOVA), controlling for organization: SUDS planning at timepoints 1, 3, and 4; Test type: Superiority; p = .43, ANCOVA

4. Secondary Outcome: Clinician Self-Efficacy Questionnaire at 4 Timepoints Across 12 Weeks
Description: Self-efficacy was measured via responses to two statements on a 7-point scale measuring clinicians' self-efficacy to use SSAIs, using established question stems from behavioral science (e.g., "If I really wanted to, I could screen every patient I see for suicide risk"). Self-efficacy was assessed separately for clinician self-efficacy for suicide screening and for use of the Safety Planning Intervention. Higher scores indicate greater self-efficacy. Scores were averaged for analysis (Range = 1 - 7).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Exposure Based Implementation Strategy (EBIS) | Implementation as Usual (IAU)
Number analyzed (Participants) | 18 | 18
units on a scale
  Time 1, screening | 5.08 (1.33) | 4.96 (1.27)
  Time 1, intervention | 4.94 (1.03) | 4.53 (1.41)
  Time 2, screening | 5.44 (1.00) | 5.06 (1.04)
  Time 2, intervention | 5.00 (1.16) | 5.22 (1.22)
  Time 3, screening: number analyzed (Participants) | 17 | 17
  Time 3, screening | 5.46 (.96) | 5.26 (1.11)
  Time 3, intervention: number analyzed (Participants) | 17 | 17
  Time 3, intervention | 5.53 (1.11) | 5.07 (1.17)
  Time 4, screening: number analyzed (Participants) | 16 | 16
  Time 4, screening | 5.75 (.91) | 5.56 (1.01)
  Time 4, intervention: number analyzed (Participants) | 16 | 16
  Time 4, intervention | 5.67 (.82) | 5.34 (1.12)
Statistical Analysis 1: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing screening self-efficacy rating at Time 3: two weeks after completing the training; Test type: Superiority; p = .59, t-test, 2 sided
Statistical Analysis 2: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing screening self-efficacy rating at Time 4: 12 weeks after completing the training; Test type: Superiority; p = .59, t-test, 2 sided
Statistical Analysis 3: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing intervening self-efficacy rating at Time 3: two weeks after completing the training; Test type: Superiority; p = .25, t-test, 2 sided
Statistical Analysis 4: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing intervening self-efficacy rating at Time 4: 12 weeks after completing the training; Test type: Superiority; p = .35, t-test, 2 sided
Statistical Analysis 5: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); repeated measures analysis of covariance (ANCOVA), controlling for organization: Self-efficacy screening at timepoints 1, 3, and 4; Test type: Superiority; p = .88, ANCOVA
Statistical Analysis 6: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); repeated measures analysis of covariance (ANCOVA), controlling for organization: Self-efficacy intervening at timepoints 1, 3, and 4; Test type: Superiority; p = .71, ANCOVA

5. Secondary Outcome: Screening Use at 3 Timepoints Across 12 Weeks
Description: Use of clinician routine suicide screening in all patient encounters was indexed via chart-stimulated recall (CSR). CSR is an established technique for examining clinician decision-making and clinical processes beyond what can be determined from chart review or self-report alone. A research team member reviewed the clinician's deidentified caseload with them for the past clinic week. For each patient seen that week, the researcher asked brief questions related to the clinicians' suicide-related practices around screening for suicide risk. Results below report the proportion of patients clinicians screened for suicide out of the total number of patients seen on one clinical day.
Time Frame: Time 1: baseline measures completed before the training; Time 3: two weeks after completing the training; Time 4: 12 weeks after completing the training
Population: This measure was completed across 3 timepoints. 2 participants dropped out of the study after post-intervention measures. 2 additional participants dropped out after two week follow up measures
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Exposure Based Implementation Strategy (EBIS) | Implementation as Usual (IAU)
Number analyzed (Participants) | 18 | 18
units
  Time 1 | .50 (.44) | .56 (.44)
  Time 3: number analyzed (Participants) | 17 | 17
  Time 3 | .49 (.46) | .52 (.35)
  Time 4: number analyzed (Participants) | 16 | 16
  Time 4 | .62 (.38) | .54 (.40)
Statistical Analysis 1: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing screening use at Time 3: two weeks after completing the training; Test type: Superiority; p = .88, t-test, 2 sided
Statistical Analysis 2: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing screening use at Time 4: 12 weeks after completing the training; Test type: Superiority; p = .55, t-test, 2 sided
Statistical Analysis 3: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); repeated measures analysis of covariance (ANCOVA), controlling for organization: CSR screening at timepoints 1, 3, and 4; Test type: Superiority; p = .36, ANCOVA

6. Secondary Outcome: Safety Planning Intervention Use (Fidelity) at Time 3 (Two Weeks After Completing the Training) and Time 4 (12 Weeks After Completing the Training)
Description: SPI Fidelity was indexed at Time 3 and Time 4 through case vignettes and standardized role play methodology. Participants received a vignette and prepare for a 45-60-minute role play, during which they were asked to complete an SPI with a patient who was determined to be at-risk for suicide following Columbia Suicide Severity Rating Scale (CSSRS) administration. Role plays were audio-recorded and coded for competence with the Safety Planning Intervention Rating Scale (SPIRS), developed by INSPIRE MPI G. Brown. This observational scale include 6 items on general safety plan intervention skills and 6 items which mapped onto the safety plan steps on a 4-point scale (0=not present to 3=excellent). Total scores were calculated by summing the 12 items with higher scores indicating greater SPI fidelity.
Time Frame: Time 3: two weeks after completing the training; Time 4: 12 weeks after completing the training
Population: This measure was completed across 2 timepoints. 2 participants dropped out after two week follow up measures
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Exposure Based Implementation Strategy (EBIS) | Implementation as Usual (IAU)
Number analyzed (Participants) | 17 | 17
score on a scale
  Time 3: total SPIRS score | 14.06 (6.71) | 11.88 (3.28)
  Time 4: total SPIRS score: number analyzed (Participants) | 16 | 16
  Time 4: total SPIRS score | 15.69 (6.65) | 15.38 (4.75)
Statistical Analysis 1: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing total SPIRS score at Time 3: two weeks after completing the training; Test type: Superiority; p = .24, t-test, 2 sided
Statistical Analysis 2: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); Test of superiority between EBIS and IAU groups comparing total SPIRS score at Time 4: 12 weeks after completing the training; Test type: Superiority; p = .88, t-test, 2 sided
Statistical Analysis 3: Comparison: Exposure Based Implementation Strategy (EBIS) vs Implementation as Usual (IAU); repeated measures analysis of covariance (ANCOVA), controlling for organization: SPIRS at timepoints 3 and 4; Test type: Superiority; p = .10, ANCOVA

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Exposure Based Implementation Strategy (EBIS) | Implementation as Usual (IAU)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-05): https://cdn.clinicaltrials.gov/large-docs/09/NCT05172609/Prot_SAP_000.pdf